CLINICAL TRIAL: NCT04031131
Title: The Use of Topical Anaesthetic in the Banding (TAB) of Internal Haemorrhoids: A Feasibility Study.
Brief Title: The Use of Topical Anaesthetic in the Banding of Internal Haemorrhoids
Acronym: TAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 258546
Record Dates: First submitted 2019-07-08; First posted 2019-07-24 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hemorrhoids
Keywords: Haemorrhoid; Banding; Topical Anaesthetic
MeSH Terms: conditions — Hemorrhoids | interventions — chlorhexidine gluconate, lidocaine drug combination

STUDY DESIGN:
Intervention Model Description: The trial will be a randomised control trial blinded to patient and assessor (the clinician collecting data at 4 hours, 72 hours and 1 month after the procedure. Randomisation will be achieved by a computer software. Administrators will be aware of which group the patient being treated is in. Half of the patients (n=30) will receive the intervention treatment (Instillagel topical anaesthetic) and lubricating gel (standard of care), the other half will receive the standard of care alone (lubricating gel) (n=30) before the procedure. The standard of care is to use no form of analgesia, with K-Y gel only being used as a lubricant. Researchers will be asked to apply the allocated treatment 5-10 minutes before the procedure. The primary end points will be: patient recruitment rate, patient acceptability, surgeon acceptability, patient retention. The secondary endpoints will be: pain scores using the 10-point visual analogue scale.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded to assessors and patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): topical anaesthetic gel and lubricating gel
  Interventions: Drug: Instillagel; Other: KY Gel
- Control Arm (Placebo Comparator): lubricating gel alone
  Interventions: Other: KY Gel

INTERVENTIONS:
Drug: Instillagel — Topical Anaesthetic Gel (Instillagel) licensed for rectal administration.
  Arms: Intervention Arm
Other: KY Gel — Lubricant Gel

SUMMARY:
The investigators' aim is to assess if they can complete a study measuring the effect of local anaesthetic gel (Instillagel) on reducing pain experienced by patients undergoing a common treatment for haemorrhoids (piles). This treatment is called rubber band ligation and is commonly performed in the investigators'clinics.

DETAILED DESCRIPTION:
A feasibility trial assessing patient recruitment, retention, randomization, and surgeon acceptability of topical anaesthetic use during rubber band ligation of haemorrhoids.

A patient and assessor blinded feasibility trial. The trial population will prospectively be recruited from colorectal surgery outpatients. Patients will be randomized to two groups to receive: lubricating gel (K-Y Jelly) and topical anaesthetic gel (Instillagel) or lubricating gel alone (the standard care).

The intervention group will receive lubricating gel and topical anaesthetic gel (containing lidocaine active ingredient) administered rectally, whilst the control group will receive lubricating gel alone (standard care). This will be carried out in Colorectal Outpatients. The band ligation of the haemorrhoids should occur between 5-10 minutes after administration of the topical anaesthetic/lubricating gel. Pain scores and the use of oral analgesia will be measured immediately after the procedure (5 minutes), upon leaving the clinic (approximately 30 minutes after), at 4 hours, and 72 hours following the procedure. Vasovagal symptoms or other complications will be recorded whilst the patient is in the clinic. At 1 month post procedure, patients will be phoned to determine if any adverse events have occurred.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic grade 1-3 haemorrhoid disease, 18+ years old, English is the first language.

Exclusion Criteria:

* Allergy to active ingredients of Instillagel, Allergy to local anaesthetic, Chronic liver disease, Grade 4 haemorrhoid disease, Pregnancy, Inflammatory bowel disease, Pre-existing anorectal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Patient recruitment rate | 5 months
  Patient recruitment rate via screening log.
Treatment acceptability to patients | 5 months
  Treatment acceptability to patients via study questionnaire. A visual analogue scale to be used, 0 - 10 with '0' being no pain and '10' being worst pain possible.
Patient retention | 5 months
  Patient retention via recruitment log.

SECONDARY OUTCOMES:
Assess if the intervention reduced pain associated with haemorrhoids up to 72 hours after the procedure, | 72 hours
  Assess if the intervention reduced pain associated with haemorrhoids up to 72 hours after the procedure via study questionnaire.
Assess if the intervention reduces vasovagal symptoms up to 72 hours after the procedure | 72 hours
  Assess if the intervention reduces vasovagal symptoms up to 72 hours after the procedure via study questionnaire.
Assess if the intervention reduced oral analgesia burden following the procedure | 72 hours
  Assess if the intervention reduced oral analgesia burden following the procedure via study questionnaire.
Assess hospital readmission 1 month after the procedure. | 1 month
  Assess hospital readmission 1 month after the procedure via review of hospital notes. The number of patients requiring additional analgesia will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Sharma, Dr, Principal Investigator — Foundation Year 1 Doctor
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson NF, Liptrott S, Maxwell-Armstrong CA. A prospective audit of early pain and patient satisfaction following out-patient band ligation of haemorrhoids. Ann R Coll Surg Engl. 2006 May;88(3):275-9. doi: 10.1308/003588406X98649. PMID 16719998
- [Background] Gokalp A, Baskonus I, Maralcan G. A prospective randomised study of local anaesthetic injection after multiple rubber band ligation of haemorrhoids. Chir Ital. 2003 Mar-Apr;55(2):213-7. PMID 12744096
- [Background] Kwok HC, Noblett SE, Murray NE, Merrie AE, Hayes JL, Bissett IP. The use of local anaesthesia in haemorrhoidal banding: a randomized controlled trial. Colorectal Dis. 2013 Apr;15(4):487-91. doi: 10.1111/codi.12088. PMID 23323626
- [Background] Law WL, Chu KW. Triple rubber band ligation for hemorrhoids: prospective, randomized trial of use of local anesthetic injection. Dis Colon Rectum. 1999 Mar;42(3):363-6. doi: 10.1007/BF02236354. PMID 10223757
- [Background] Hooker GD, Plewes EA, Rajgopal C, Taylor BM. Local injection of bupivacaine after rubber band ligation of hemorrhoids: prospective, randomized study. Dis Colon Rectum. 1999 Feb;42(2):174-9. doi: 10.1007/BF02237123. PMID 10211492